CLINICAL TRIAL: NCT03506451
Title: PaRTNer: Patient Reported Outcomes and Financial Toxicity in Head and Neck Cancer A Pilot, Survey Based Study
Acronym: PaRTNer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00092590
Record Dates: First submitted 2018-04-20; First posted 2018-04-24 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Cancer
Keywords: Financial toxicity
MeSH Terms: conditions — Head and Neck Neoplasms; Financial Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm non-therapeutic interventional study (Other): All subjects who enroll on study will be asked to complete questionnaires at baseline before treatment starts; the questionnaires are repeated at one month, three and six months after radiation therapy has been completed. the demographics questionnaire is completed at baseline only; the FACT-HN is completed at all four time points.
  Interventions: Other: Demographics questionnaires and the FACT HN questionnaire

INTERVENTIONS:
Other: Demographics questionnaires and the FACT HN questionnaire — Patients will complete a baseline survey assessing socioeconomic household information, baseline symptoms, QOL, and financial toxicity, as well as attitudes toward cost conversations and educational handouts.

SUMMARY:
The purpose of this single institution, pilot study is to explore the out of pocket (OOP)costs and financial toxicity of cancer care for patients during definitive treatment of head and neck cancer with radiation therapy with or without chemotherapy and surgical resection. The study team will assess how the financial burden of cancer care impacts quality of life as well as treatment-related decision-making from a patient perspective.

DETAILED DESCRIPTION:
This is a prospective, single institution, survey-based study to assess OOP costs, financial toxicity and pateint reported outcomes (PROs') (including QOL, quality of care, and attitudes/perspectives on the role of cost in treatment decisions). Potential participants are new patient consults in Radiation Oncology Head and Neck Cancer Clinic. Patients with an indication for definitive treatment involving radiation therapy will be approached by study staff and, if amenable, enrolled in the study. After signing informed consent, they will complete a baseline survey assessing socioeconomic household information, baseline symptoms/QOL and baseline costs/financial toxicity. They will be followed prospectively and re-surveyed at 3 and 6 months after completion of radiation therapy. Repeat assessments will document treatment costs and PRO including QOL, financial toxicity, and self-reported quality of care. Patients will be asked to collect all treatment-related bills in a provided binder, which will be reviewed at each survey date. Basic demographic data (including age, sex, race, marital status, zip code, and insurance coverage), comorbidities, smoking status, cancer characteristics (stage, site, histology), treatments received, emergency department visits and hospitalization rates at baseline, end of treatment, 3 months and 6 months after radiation treatment will be collected as part of this study. Disease status and survival will also be assessed from standard of care follow-up visits up to five years after completion of radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (18 years or older) patients
2. Diagnosed with HNC with treatment plan including definitive radiation therapy or chemotherapy/radiation therapy
3. Be able to read and write in English
4. Able to give informed consent and complete survey materials

Exclusion Criteria:

1. Recurrent disease
2. Metastatic disease
3. Prior radiation courses must be approved by PI prior to approaching patient for enrollment (prior systemic therapy is not an exclusion to study enrollment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2026-10-07 (Estimated)

PRIMARY OUTCOMES:
Financial toxicity, as measured by out of pocket (OOP) costs for a definitive course of treatment for HNC | 3 months post radiation therapy
Financial toxicity, as measured by out of pocket (OOP) costs for a definitive course of treatment for HNC | 6 months post radiation therapy
Financial toxicity, as measured by change in Comprehensive Score for financial Toxicity (COST) | Baseline, 3 months post radiation therapy, 6 months post radiation therapy
  Financial toxicity will be measured using the comprehensive score for financial toxicity (COST). The range of the COST score is 0-44.

SECONDARY OUTCOMES:
Change in symptom burden, as measured by Functional Assessment of Cancer Therapy-Head and Neck (FACT-H&N) score | Baseline, 3 months post radiation therapy, 6 months post radiation therapy
Change in quality of life, as measured by FACT-H&N score | Baseline, 3 months post radiation therapy, 6 months post radiation therapy
Perceived quality of care | 3 months post radiation therapy, 6 months post radiation therapy
  Patients will be asked to rate the quality of care as excellent, good, fair, poor, or very poor

OTHER OUTCOMES:
Disease status | 5 years post completion of radiation treatment
Overall survival | 5 years post completion of radiation treatment
Progression free survival | 5 years post completion of radiation treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Karukonda, MD, Principal Investigator — Duke University Health System (DUHS)
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No